CLINICAL TRIAL: NCT05682898
Title: Perioperative Management of Colorectal Cancer Patients Infected With COVID-19: a Multicenter Prospective Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Professor, Changhai Hospital
Other Study IDs: WeiZhang
Record Dates: First submitted 2023-01-11; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Surgical Procedure, Unspecified
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- More than 7 weeks: Timing of colorectal cancer surgery is more than 7 weeks after confirmed COVID-19 infection by COVID-19 nucleic acid test.
  Interventions: Procedure: Timing of colorectal cancer surgery
- Less than 7 weeks: Timing of colorectal cancer surgery is less than 7 weeks after confirmed COVID-19 infection by COVID-19 nucleic acid test.
  Interventions: Procedure: Timing of colorectal cancer surgery

INTERVENTIONS:
Procedure: Timing of colorectal cancer surgery — The timing of colorectal cancer surgery is different according patients' different conditions which is difined as more than 7 weeks or less than 7 weeks.

SUMMARY:
This trial is a multicenter prospective cohort study to explore timing of colorectal cancer surgery after COVID-19 infection so that can assist clinicians and patients. Currently, there is less evidence on perioperative outcomes after COVID-19 vaccination and the omicron variant. Therefore, it is necessary to update previously published consensus which recommends that patients should avoid elective surgery within 7 weeks of COVID-19 infection remain, unless the benefits of doing so exceed the risk of waiting. Aiming at the above problems, we plan to carry out a multicenter prospective cohort study to develop perioperative management according patients' different conditions.

ELIGIBILITY:
Inclusion Criteria:

* undergoing colorectal cancer surgery
* infected with COVID-19 but nucleic acid test result is negative
* the patients compliance is good
* signed the consents voluntarily

Exclusion Criteria:

* undergoing emergency surgery(intestinal obstruction, intestinal perforation, intestinal hemorrhage, et al.)
* The patients' situations which judged by situations is not suitable to participate in the clinical trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Colorectal cancer patients undergoing surgery with perioperative COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical complications | 30 days after surgery
  Complications including: intraperitoneal hemorrhage, anastomotic leak, anastomotic bleeding, abdominal infection, pulmonary infection, chylous fistula, intestinal obstruction, et al.